CLINICAL TRIAL: NCT04441944
Title: TELEmedicine as an Intervention for Sepsis in Emergency Departments
Acronym: TELEvISED
Status: Completed | Type: Observational
Sponsor: University of Iowa (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Nicholas M Mohr, Professor, University of Iowa
Other Study IDs: 201901748
Record Dates: First submitted 2020-06-17; First posted 2020-06-22 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Sepsis
Keywords: Telemedicine
MeSH Terms: conditions — Sepsis | interventions — Telemedicine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Telemedicine Cases: Patients presenting to rural emergency departments who had real-time provider-to-provider telemedicine used to supplement their emergency department care.
  Interventions: Other: Telemedicine
- Non-Telemedicine Cases: Patients presenting to rural emergency departments who did not have real-time provider-to-provider telemedicine used to supplement their emergency department care.

INTERVENTIONS:
Other: Telemedicine — Use of provider-to-provider telemedicine
  Groups: Telemedicine Cases

SUMMARY:
Sepsis is a life-threatening condition that has doubled in incidence over the past decade, and timely aggressive medical intervention has been shown to save lives. Rural sepsis patients have a 38% higher mortality rate, possibly attributable to delays in early sepsis care. Rural emergency department (ED)-based provider-to-provider telemedicine has been proposed to standardize care and support local clinicians in rural hospitals. The goal of this multicenter observational comparative effectiveness study is to measure the association between tele-ED use and clinical outcomes in a cohort of rural sepsis patients.

DETAILED DESCRIPTION:
Sepsis is a life-threatening condition that has doubled in incidence over the past decade, and timely aggressive medical intervention has been shown to save lives. Rural sepsis patients have a 38% higher mortality rate, possibly attributable to delays in early sepsis care. This effect persists even among patients who are transferred between hospitals and who bypass rural hospitals. With 17% of all hospital deaths attributable to sepsis and 19% of Americans living in rural areas, there is a critical need to identify strategies to reduce the disparities in outcomes between rural and urban sepsis care.

Rural ED-based telemedicine has been proposed to standardize care and support local clinicians in rural hospitals. Telemedicine networks provide a real-time, high-definition on-demand video connection between a rural hospital and a tertiary hub 24 h daily. Based in Sioux Falls, South Dakota, Avera eCare is a tele-emergency network that serves as a hub for a 140-hospital network that spans 12 rural Midwestern states. It is the largest rural ED-based telehealth network in North America, and a network the investigators have studied previously.

Our central hypothesis is that telemedicine will improve clinical outcomes through improved adherence with Surviving Sepsis Campaign (SSC) guidelines. Using comparative effectiveness methods and a patient-centered outcomes research (PCOR) approach, this study will test the hypotheses with the following specific aims:

1. To measure the association between rural ED-based telemedicine use, guideline adherence, and clinical outcomes using an observational cohort comparative effectiveness research study. Rural clinicians choose whether individual sepsis patients will be treated with telemedicine-supplemented care. Medical records will be analyzed from patients with severe sepsis who present to 25 rural hospital EDs that are part of a telemedicine network to estimate the effect of telemedicine on changing early SSC guideline adherence. Guideline adherence has been studied extensively as an outcome of sepsis implementation studies. The study will also analyze the impact of telemedicine on clinical outcomes, such as mechanical ventilation, hospital length-of-stay, and survival, using mediation analysis in a propensity-matched cohort design. Our working hypothesis is that telemedicine consultation will improve SSC guideline adherence and will reduce delays in care, leading to improved clinical outcomes.
2. To measure the effect of ED-based telemedicine on guideline adherence among patients who have telemedicine available but not used. In addition to the effect of use for individual patient care, telemedicine interactions may provide ongoing training for providers and nurses and influence care even for patients for whom telemedicine is not used. This effect may result from a learning effect in which local providers adopt practices they observe in telemedicine-consulted patients. The investigators will use hospital fixed-effects models to measure this association. The working hypothesis is that guideline adherence will increase after telemedicine adoption even in non-telemedicine patients, and adherence will be associated with the number of prior telemedicine sepsis encounters (dose-response).

The rationale for this research is that dissemination and implementation of best practices through rural networks remains difficult, but telemedicine offers one potential solution. Sepsis is an ideal model to study the effect of telemedicine because it differs from other acute care conditions treated in rural hospitals (e.g., trauma, myocardial infarction) in that early treatment provided in rural hospitals may be more important than rapid transfer to tertiary centers. Focusing on telemedicine in rural sepsis care will serve as a powerful model for examining strategies for disseminating innovations across rural networks.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age 18 years or older)
* Arrive at participating emergency department between August 1, 2016 and June 30, 2019
* Hospital diagnosis of infection and organ failure
* Identification of infection in the emergency department
* Presence of organ failure in the emergency department (SOFA score of at least 2)
* Presence of systemic inflammatory response syndrome (SIRS) in the emergency department

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study will include all adult (age≥18 years) sepsis patients who presented to a participating rural ED between August 1, 2016 and June 30, 2019. Because of poor sensitivity in diagnosis code-based definitions of sepsis, we elected to use a multi-step definition requiring (1) hospital diagnosis of both infection and organ failure, (2) identification of infection in the ED, (3) presence of organ failure in the ED, and (4) presence of systemic inflammatory response syndrome (SIRS) criteria in the ED. To identify hospital diagnosis of infection and organ failure, we used the Fleischmann-Struzek approximation of sepsis using International Classification of Diseases, 10th edition, Clinical Modification (ICD-10-CM) or an explicit sepsis code (R65.20 or R65.21).
Sampling Method: Probability Sample
Enrollment: 1191 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
28-day Hospital-Free Days | Within 28 days of emergency department presentation
  The total number of days in the 28 days after emergency department presentation that a patient is alive and outside the hospital.

SECONDARY OUTCOMES:
Surviving Sepsis Campaign Guideline Adherence | 6 hours after emergency department arrival
  Adherence with all elements of the Surviving Sepsis Campaign 3-hour and 6-hour bundles (dichotomous)
Mortality | Through hospital discharge, an average of 8 days
  Did patient die in the hospital?
Mechanical Ventilation | Through hospital discharge, an average of 8 days
  Was mechanical ventilation required during admission?
Vasopressors | Through hospital discharge, an average of 8 days
  Was vasopressor therapy required during admission?
New Hemodialysis | Through hospital discharge, an average of 8 days
  Was dialysis required during this admission (if not on chronic dialysis)?
Inter-hospital Transfer | Through hospital discharge, an average of 8 days
  Was inter-hospital transfer required from the index hospital?
28-Day Ventilator-Free Days | 28 days
  The total number of days in the 28 days after emergency department presentation that a patient is alive and not requiring a ventilator.
28-Day Vasopressor-Free Days | 28 days
  The total number of days in the 28 days after emergency department presentation that a patient is alive and not requiring a vasopressor.
28-Day ICU-Free Days | 28 days
  The total number of days in the 28 days after emergency department presentation that a patient is alive and not requiring an ICU bed.
Emergency Department Length-of-Stay | Index emergency department duration (1 day)
  The total duration of stay in the index emergency department.
Time-to-inpatient unit arrival | 24 hours
  The time from index emergency department registration to arrival in the inpatient unit

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Mohr, MD, MS, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No
Aggregate data will be shared with investigators who make a written request to the study team. These data will include aggregate effect sizes, but will not be patient-level data. Because of the sparsely populated region where this study is being conducted, hospital-identifiable data would be sufficient to identify individuals in this region, so fully de-identifying this data set would make it unusable for subsequent independent analyses (e.g., would require removing age, sex, hospital, transfer distance, transport times, comorbidities). The study team will, however, collaborate with other investigators to conduct additional analysis, maintaining the security of the data set.

REFERENCES:
- [Derived] Mohr NM, Okoro U, Harland KK, Fuller BM, Campbell K, Swanson MB, Wymore C, Faine B, Zepeski A, Parker EA, Mack L, Bell A, DeJong K, Mueller K, Chrischilles E, Carpenter CR, Wallace K, Jones MP, Ward MM. Outcomes Associated With Rural Emergency Department Provider-to-Provider Telehealth for Sepsis Care: A Multicenter Cohort Study. Ann Emerg Med. 2023 Jan;81(1):1-13. doi: 10.1016/j.annemergmed.2022.07.024. Epub 2022 Oct 15. PMID 36253295
- [Derived] Mohr NM, Harland KK, Okoro UE, Fuller BM, Campbell K, Swanson MB, Simpson SQ, Parker EA, Mack LJ, Bell A, DeJong K, Faine B, Zepeski A, Mueller K, Chrischilles E, Carpenter CR, Jones MP, Ward MM. TELEmedicine as an intervention for sepsis in emergency departments: a multicenter, comparative effectiveness study (TELEvISED Study). J Comp Eff Res. 2021 Feb;10(2):77-91. doi: 10.2217/cer-2020-0141. Epub 2021 Jan 20. PMID 33470848